CLINICAL TRIAL: NCT00274755
Title: Improved Characterization of Brain Tumors By MRI and MRS
Brief Title: Magnetic Resonance Imaging and Magnetic Resonance Spectroscopic Imaging in Evaluating Patients Who Are Undergoing Treatment for Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000441015; UCSF-05106
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult diffuse astrocytoma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult pilocytic astrocytoma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Glioblastoma; Gliosarcoma; Ependymoma; Glioma, Subependymal; Oligodendroglioma; Glioma | interventions — Drug Therapy; Magnetic Resonance Spectroscopy; Radiotherapy

INTERVENTIONS:
Drug: chemotherapy
Procedure: conventional surgery
Procedure: magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging
Radiation: radiation therapy

SUMMARY:
RATIONALE: Diagnostic procedures, such as magnetic resonance imaging (MRI) and magnetic resonance spectroscopic imaging (MRSI), (done before, during, and after treatment) may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase II trial is studying how well MRI and MRSI evaluate patients who are undergoing treatment for gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the magnetic resonance spectroscopic imaging (MRSI) characteristics of patients who are undergoing treatment for supratentorial glioma.
* Determine the survival of patients who undergo magnetic resonance imaging and MRSI.
* Determine the clinical outcome of patients who undergo these imaging procedures.
* Correlate measures of metabolic tumor burden (i.e., CNI, CCCrI, CrNI, and LLI) with survival and clinical outcome in patients who undergo these imaging procedures.
* Determine the time to clinical progression in patients who undergo these imaging procedures.

OUTLINE: Patients are assigned to 1 of 2 treatment groups based on grade of disease.

* Group 1 (patients with grade II glioma): Patients undergo magnetic resonance imaging (MRI) and magnetic resonance spectroscopic imaging (MRSI). Patients then receive chemotherapy. Patients undergo repeat MRI/MRSI after courses 2 and 4 of chemotherapy.
* Group 2 (patients with grade III-IV glioma): Patients undergo MRI/MRSI and then undergo surgical resection of the tumor. Patients then receive chemoradiotherapy. Patients undergo repeat MRI/MRSI within 2 weeks and at 2 months after completion of radiotherapy.

Patients are followed for recurrence, disease progression, and survival.

PROJECTED ACCRUAL: A total of 250 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial glioma

  * Grade II-IV disease
  * Previously untreated disease
* Eligible for surgical resection and/or chemotherapy with or without radiotherapy
* Tumor accessible by magnetic resonance spectroscopic imaging

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 8 weeks
* Not pregnant
* No contraindication for magnetic resonance examinations, including any of the following:

  * Cardiac pacemaker or fibrillator
  * Aneurysm clip
  * Insulin or infusion pump
  * Any implant held in place by a magnet
  * Metal contamination anywhere in the body

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior radiotherapy
* No prior treatment for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2003-11; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Survival
Time to clinical progression

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J. Nelson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States